CLINICAL TRIAL: NCT03484052
Title: Place of Jugular Ultrasound in the Evaluation of the Volemia by a Clinician Doctor in Routine Care (JUVIA)
Brief Title: Place of Jugular Ultrasound in the Evaluation of the Volemia by a Clinician Doctor in Routine Care
Acronym: JUVIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC17_8832_JUVIA
Record Dates: First submitted 2018-03-16; First posted 2018-03-30 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jugular ultrasound (Other)
  Interventions: Other: Jugular ultrasound

INTERVENTIONS:
Other: Jugular ultrasound — Performing a jugular ultrasound by 2 operators before and after transfusion

SUMMARY:
Interventional study with minimal risks and constraints, prospective, monocentric.

DETAILED DESCRIPTION:
To appreciate the volemia of a patient is a frequent problem in hospital in various situations: renal insufficiency, dyspnea, dysnatremia, etc. The aging of the population, the chronicity of pathologies, overweight among other causes can make it difficult to assess the volume of the disease by the clinic alone. The consequences of a poor evaluation are delayed management and possible iatrogeny.

New discrimination markers have emerged to help the clinician such as "brain natriuretic peptide (BNP)" in dyspnea, and especially transthoracic echocardiography (TTE) assessing filling pressures with a high potency. discrimination. In current practice the TTE has unequal accessibility, and requires trained practitioners. It is difficult to have an TTE performed for all patients where the question arises.

Just as an assessment of the initial volemia is often necessary, there are few objective monitoring criteria. One can quote the variation of the weight or the evolution of certain biological parameters but none is completely specific.

A new marker has been described for a few years: jugular ultrasound. Better accessibility (requires only a probe of 7-9Hz, possibly 5Hz), it can indeed be performed by any practitioner in less than a minute. The jugular distension is a reflection of cardiac pre-load and can be correctly estimated by ultrasound. It has been shown that cardiac decompensated patients have dilated jugular veins compared to a reference population. A low cohort also demonstrated the presence of jugular ultrasound distension in the absence of clinical distension.

In a US study, 119 patients admitted to the emergency department for dyspnea had a sensitivity of 99% for a specificity of 59% for trans-jugular ultrasound in cardiogenic edema.

However, many applications remain to be explored, and the repeated use of jugular ultrasound in the same patient has never been studied. The accessibility of the measure could make it an excellent monitoring tool.

As a clinical situation, the investigators chose a well standardized and studied situation such as blood transfusion that can bridge the preload measured by invasive measures and measured by jugular ultrasound. This situation is complicated in patients in 1 to 5.7% of the situations of secondary pulmonary overload.

ELIGIBILITY:
Inclusion Criteria:

* Major patient;
* Requiring a transfusion of 2 or more red blood cells in a routine care situation (transfusion programmed in the context of a day hospital or a traditional hospitalization, except in cases of massive bleeding);
* Affiliate or beneficiary of a social protection scheme;
* Having given his written consent.

Exclusion Criteria:

* Patient with clinical or biological criteria for admission to intensive care as defined in the 1999 US ICU Practice Guidelines;
* Major persons subject to legal protection (legal safeguards, guardianship, tutorship), persons deprived of their liberty;
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of the volemia | Baseline
  Variation in height of the area where the right jugular vein collapses in centimeters from the angle of Louis.

SECONDARY OUTCOMES:
Transfusion tolerance | Day 3
  Study of transfusion tolerance (pre- and post-transfusion clinical collection, oral interview on D3 with the patient).
Interobserver variability | Baseline
  Inter-observer variability evaluated by the Intra-class Correlation Coefficient
Interobserver variability | Baseline
  Inter-observer variability evaluated by the Bland and Altman graph.
Semi-quantitative measurement variation in the height of the zone where the right jugular vein colludes | Baseline
  The semi-quantitative variation in height measurement will be evaluated by a Chi² test or an exact Fisher test in two ways: improvement observed or no improvement observed

CONTACTS AND LOCATIONS:
Overall Officials: JEGO Patrick, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Britain, France

REFERENCES:
- [Result] Henriot B, Scanff A, Sebillot M, Lautredoux F, Jego P. Jugular vein ultrasound for estimating changes in blood volume: a new tool for all physicians. Intern Emerg Med. 2021 Oct;16(7):2005-2007. doi: 10.1007/s11739-021-02792-y. Epub 2021 Jul 1. No abstract available. PMID 34196887